CLINICAL TRIAL: NCT01954888
Title: Impact of the Ultrasound-guided Approach on the Efficiency and Safety of the Stellate Ganglion Block in Chronic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Veronique Brulotte, Impact of the ultrasound-guided approach on the efficiency and safety of the stellate ganglion block in chronic pain, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13054
Record Dates: First submitted 2013-09-26; First posted 2013-10-07 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blind technique (Active Comparator): Stellate ganglion block using the anterior paratracheal approach using surface landmarks.
  Interventions: Procedure: Blind technique
- Ultrasound-guided technique (Active Comparator): Stellate ganglion block using the ultrasound-guided lateral approach at the sixth cervical vertebral level.
  Interventions: Procedure: Ultrasound-guided technique

INTERVENTIONS:
Procedure: Blind technique — A mixture of 3 mL of 2% lidocaine and 7 mL of 0.5% bupivacaine is used for both approaches (blind and ultrasound-guided).
  Arms: Blind technique
Procedure: Ultrasound-guided technique — A mixture of 3 mL of 2% lidocaine and 7 mL of 0.5% bupivacaine is used for both approach (blind and ultrasound-guided).
  Arms: Ultrasound-guided technique

SUMMARY:
The first purpose of this study is to compare the effectiveness of the stellate ganglion block realized with two different approaches (blind and ultrasound-guided) in patients with a diagnosis of complex regional pain syndrome.

The second purpose of this study is to determine the safest approach and to compare the safety profiles of the two approaches.

DETAILED DESCRIPTION:
To evaluate whether the ultrasound guided approach is more effective than the blind technique in producing a greater than 1.5 degree Celsius rise in ipsilateral arm temperature after a stellate ganglion block.

Blocks will both be performed with 10 mL of xylocaine/bupivacaine. Secondary outcomes will be the impact of the approach (blind vs ultrasound) on pain reduction, horner syndrome, side effects (hoarseness, dysphagia, pharyngeal discomfort) and complications (blood aspiration, intravascular injection).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years
* Patients with a new or known diagnosis of complex regional pain syndrome (according to the criteria of Budapest) at the upper extremity

Exclusion Criteria:

* Refusal of a patient
* Coagulopathy
* Systemic infection or local infection at the needle injection site
* Major deformation at the level of the neck (radiotherapy, surgery, etc. )
* Concomitant chronic pain syndrome
* Post-pneumonectomy on the controlateral side
* Severe hepatic impairment or severe renal impairment (Clcr under 30 ml/min)
* Known allergy to local anesthetics of amide type
* Inability to understand a numeric pain scale

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-09; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
proportion of patients reaching >1.5 °C rise in ipsilateral arm temperature | thirty minutes after block

SECONDARY OUTCOMES:
Complications | Time of the block to one week after the block
  Seizure, loss of consciousness with apnea, hematoma, recurrent laryngeal nerve injury, phrenic nerve paralysis, pneumothorax, weakness of the ipsilateral upper limb, foreign body sensation

OTHER OUTCOMES:
Severity of pain | Immediately and each day after the block until one week after the block
  The severity of the pain will be evaluated before the block and each day after the block for one week using a numeric rating scale (0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Brulotte, MD, MSC, FRCPC, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhatia A, Flamer D, Peng PW. Evaluation of sonoanatomy relevant to performing stellate ganglion blocks using anterior and lateral simulated approaches: an observational study. Can J Anaesth. 2012 Nov;59(11):1040-7. doi: 10.1007/s12630-012-9779-4. Epub 2012 Sep 6. PMID 22956268